CLINICAL TRIAL: NCT06200467
Title: A Double-blind, Randomized, Placebo-controlled, Multiple-dose, Parallel Group With Nested Crossover Design Trial With Moxifloxacin as Positive Control to Evaluate the Effects of Multiple Subcutaneous Doses of BI 456906 in a Titration Scheme on Cardiac Safety Parameters in (Otherwise) Healthy Male and Female Subjects With Overweight/Obesity
Brief Title: A Study to Test Whether Multiple Doses of BI 456906 Have an Effect on Cardiac Safety in People With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1404-0011; 2023-506375-10-00 (Registry Identifier: CTIS); U1111-1295-4369 (Other: WHO Registry)
Record Dates: First submitted 2023-12-28; First posted 2024-01-11 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — BI 456906; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Parallel group design trial, with moxifloxacin as positive control in a nested cross-over in healthy male and female subjects with overweight/obesity.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm A: R1 then R3 then T then R (Experimental): Arm A: BI 456906-placebo (reference treatment 1 (R1)) then moxifloxacin-placebo (reference treatment 3 (R3)) then BI 456906 (Test Treatment (T)) then moxifloxacin-placebo (R3)
  Interventions: Drug: BI 456906; Drug: Placebo to BI 456906; Drug: Placebo to moxifloxacin
- Arm B: R1 then R2 then R1 then R3 (Placebo Comparator): Arm B: BI 456906-placebo (R1) then moxifloxacin (Reference Treatment 2 (R2)) then BI 456906-placebo (R1) then moxifloxacin-placebo (R3)
  Interventions: Drug: Placebo to BI 456906; Drug: Moxifloxacin; Drug: Placebo to moxifloxacin
- Arm C: R1 then R3 then R1 then R2 (Placebo Comparator): Arm C: BI 456906-placebo (R1) then moxifloxacin-placebo (R3) then BI 456906-placebo (R1) then moxifloxacin (R2)
  Interventions: Drug: Placebo to BI 456906; Drug: Moxifloxacin; Drug: Placebo to moxifloxacin

INTERVENTIONS:
Drug: BI 456906 — Solution for injection
  Other Names: survodutide
  Arms: Arm A: R1 then R3 then T then R
Drug: Placebo to BI 456906 — Solution for injection
  Other Names: BI 456906-placebo
Drug: Moxifloxacin — Film-coated tablet
  Arms: Arm B: R1 then R2 then R1 then R3; Arm C: R1 then R3 then R1 then R2
Drug: Placebo to moxifloxacin — Film-coated tablet

SUMMARY:
This study is open to adults between 18 and 55 years of age with overweight or obesity. The purpose of this study is to find out whether a medicine called survodutide (BI 456906) has an effect on cardiac safety. When a new medicine is developed, it is important to check whether it affects the heart. Moxifloxacin is a medicine that is known to change the heart rhythm. In this study, moxifloxacin is used as a so-called positive control.

Participants are put into 3 groups by chance. There is a different treatment schedule for each of the groups. All participants start with one placebo injection under their skin. The next day, depending on the group, participants take either moxifloxacin or placebo as a tablet. Then, for about 30 weeks, participants receive survodutide or placebo as an injection under their skin once a week. After this, they take again a single dose of moxifloxacin or placebo.

Participants are in the study for up to 9 months. During this time, they visit the study site regularly. For 2 of the visits, participants stay at the study site for 2 nights. During these visits, the doctors collect information about participants' health. To assess the study endpoints, the study staff regularly performs ECG tests. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 55 years (inclusive)
3. Body mass index (BMI) of 27.0 to 39.9 kg/m2 (inclusive) and body weight > 70 kg
4. Signed and dated written informed consent in accordance with the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
5. Female subjects who meet any of the following criteria for a highly effective contraception from at least 7 days before the first administration of trial medication until 28 days after trial completion:

   * Use of combined (estrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal or transdermal). In case of oral contraception a barrier method should be used in addition.
   * Use of progestogen-only hormonal contraception that inhibits ovulation (oral, injectable or implantable). In case of oral contraception a barrier method should be used in addition.
   * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
   * Sexually abstinent
   * A vasectomised sexual partner who received medical assessment of the surgical success (documented absence of sperm) and provided that partner is the sole sexual partner of the trial participant
   * Surgically sterilised (including hysterectomy)
   * Postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of Follicle Stimulating Hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance and, in particular:

   * Alanine aminotransferase (ALT) above upper limit of normal (ULN) + 20%
   * Aspartate aminotransferase (AST) above ULN + 20%
   * Gamma glutamyltransferase (GGT) above ULN + 20%
   * Lipase or amylase above ULN + 20%
   * Bilirubin above 1.2x ULN (except for cases of Gilbert's Syndrome)
   * eGFR < 60 mL/min/1.73 m²
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. History of either chronic or acute pancreatitis
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Time-matched QTcI change from baseline (ΔQTcI) collected at the same time points as the BI 456906 plasma concentrations up to a maximum of 30 weeks after first drug administration of BI 456906 / BI 456906-placebo | up to 30 weeks.
  QTcI is the QT interval (electrocardiogram interval from the start of the QRS complex (combination of the Q wave, R wave and S wave) to the end of the T wave) individually corrected for heart rate.

SECONDARY OUTCOMES:
The QTcI change from baseline (ΔQTcI) collected at the same time points as the moxifloxacin plasma concentrations up to 12 hours after drug administration of a single dose of moxifloxacin or moxifloxacin-placebo | up to 12 hours.
The time-matched heart rate change from baseline (ΔHR) collected at the same time points as the BI 456906 plasma concentrations up to a maximum of 30 weeks after first drug administration of BI 456906 / BI 456906-placebo | up to 30 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com